CLINICAL TRIAL: NCT02100631
Title: A Phase III Randomized, Double-blind, Placebo-controlled Study in Older Adults to Assess Immunogenicity and Clinical Acceptability of a Single-dose of the Live Oral Cholera Vaccine Candidate PXVX0200 O1 Serotype Inaba Strain CVD 103-HgR
Brief Title: A Study of Live Oral Cholera Vaccine, PXVX200 in Healthy Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PXVX-VC-200-005
Record Dates: First submitted 2014-03-25; First posted 2014-04-01 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PXVX0200 in Older Adults (Experimental): PXVX0200 Single dose; liquid suspension after reconstitution with buffer; > 2x10^8 CFU in a liquid suspension
  Interventions: Biological: PXVX0200
- Placebo in Older Adults (Placebo Comparator): Placebo physiological saline
  Interventions: Biological: Placebo
- Historical Control: Adults Aged 18-45 (Other): This arm consists of historical data from subjects who received a single dose of PXVX0200 in study PXVX-VC-200-004. The data was included in study PXVX-VC-200-005 as a comparator bridging population for the Day 11 seroconversion. NCT02094586 PubMed ID:29317118
  Interventions: Biological: PXVX0200

INTERVENTIONS:
Biological: PXVX0200
  Arms: Historical Control: Adults Aged 18-45; PXVX0200 in Older Adults
Biological: Placebo
  Arms: Placebo in Older Adults

SUMMARY:
Demonstrate that the vaccine offers protection based on antibody levels in older adults and is similar to antibody levels in adults aged 18-45 following vaccination with PXVX0200.

DETAILED DESCRIPTION:
Demonstrate that seroconversion by classical Inaba vibriocidal antibody at Day 11 in older adults ages 46-64 years (inclusive) was non inferior to seroconversion at Day 11 in younger adults ages 18-45 years following vaccination with PXVX0200.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and give written consent.
2. Healthy male and female adults, age 46-64 years (inclusive) without significant medical history, physical, or abnormal screening laboratory test results at screening.
3. Women of childbearing potential must have had a negative urine pregnancy test at screening, prior to vaccination. Female subjects must be of non-childbearing potential (as defined as surgically sterile or postmenopausal for more than 1 year), or if of childbearing potential must be practicing abstinence or using an effective licensed method of birth control (eg, use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, intrauterine devices [IUDs], cervical sponges, diaphragms, condoms with spermicidal agents; or must have a vasectomized partner) within 2 months of vaccination and must agree to continue such precautions during the study.
4. Willing and able to comply with the study requirements and procedures.

Exclusion Criteria:

1. Currently active unstable or undiagnosed medical conditions including immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurologic illness, psychiatric disorder requiring hospitalization, current drug or alcohol abuse. Examples of unstable or undiagnosed medical conditions including unstable angina pectoris, shortness of breath on exertion without clear etiology and chronic renal failure requiring dialysis. Examples of conditions that do not meet exclusion criteria include mild controlled hypertension, mild controlled asthma, and treated depression without hospitalization.
2. Abnormal stool pattern defined as fewer than 3 stools per week or more than 2 stools per day in past 6 months.
3. Regular use of laxatives in the past 6 months.
4. Previously received a licensed or investigational cholera vaccine.
5. History of cholera or enterotoxigenic E. coli infection (natural infection or experimental challenge).
6. Travel to a cholera-endemic area in the previous 5 years.
7. Received or plans to receive any other licensed vaccines, except for seasonal influenza vaccine, from 14 days prior to the study vaccination through to 29 days after vaccination.
8. Received or plans to receive antibiotics or chloroquine within 14 days prior to the study vaccination through to 29 days after vaccination.
9. Recipient of bone marrow or solid organ transplant.
10. Use of systemic chemotherapy in the previous 5 years prior to the study.
11. Malignancy (excluding non-melanotic skin cancers) or lymphoproliferative disorders diagnosed or treated during the past 5 years.
12. Received or plans to receive systemic immunosuppressive therapy, radiation therapy, parenteral or high-dosage inhaled steroids (>800 µg/day of beclomethasone diproprionate or equivalent) within 6 months prior to the study vaccination through to Day 29.
13. History of Guillain-Barré Syndrome.
14. Pregnant or nursing.

Ages: 46 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 398 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarty, MD, Study Director — Emergent Travel Health Inc.
Locations (16):
- United States (16):
  - Coastal Clinical Research, Mobile, Alabama
  - Avail Clinical, DeLand, Florida
  - Miami Research Associates, Miami, Florida
  - Palm Beach Research Center, Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Heartland Research, Wichita, Kansas
  - Central Kentucky Research, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Boston University, Boston, Massachusetts
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Research Across America, Dallas, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCarty JM, Lock MD, Bennett S, Hunt KM, Simon JK, Gurwith M. Age-related immunogenicity and reactogenicity of live oral cholera vaccine CVD 103-HgR in a randomized, controlled clinical trial. Vaccine. 2019 Mar 7;37(11):1389-1397. doi: 10.1016/j.vaccine.2019.01.077. Epub 2019 Feb 13. PMID 30772070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included healthy volunteers (46 - 64 years) who were not previously immunized against cholera. A total of 398 subjects randomized, of which 299 received study treatment and 99 received placebo. A total of 36 subjects from the treatment group continued in the Immune Sub-study population.
Pre-assignment Details: This study included healthy volunteers (46 - 64 years) who were not previously immunized against cholera. A total of 398 subjects randomized, of which 299 received study treatment and 99 received placebo. A total of 36 subjects from the treatment group continued in the Immune Sub-study population.
  The historical control subjects are not included in the protocol enrollment number for PXVX-VC-200-005. They are solely a comparator population.
Groups:
- PXVX0200 in Older Adults: PXVX0200 Single dose; liquid suspension after reconstitution with buffer; > 1x10^9 CFU in a liquid suspension
Period: Overall Study
Arm/Group | PXVX0200 in Older Adults | Placebo in Older Adults | Historical Control: Adults Aged 18-45
Started | 299 | 99 | 2688
Completed | 292 | 95 | 2688
Not Completed | 7 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0
Not completed — 3 subjects randomized to treatment unable to receive vaccine as product not available, | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PXVX0200 in Older Adults: PXVX0200 is a live-attenuated cholera vaccine for single-dose oral administration. Subjects will be randomly assigned 3:1 to receive PXVX0200 (300) or placebo (100). Each subject will have at least 4 visits composed of a screening visit, a vaccination visit (Day 1), and post-vaccination visits at Day 11, and Day 29 telephone contacts will be made on Day 91 and 181.
- Placebo in Older Adults: The placebo consisted of 100 mL of physiological saline administered orally. Physiological saline was sourced by the clinical sites. Subjects will be randomly assigned 3:1 to receive PXVX0200 (300) or placebo (100). Each subject will have at least 4 visits composed of a screening visit, a vaccination visit (Day 1), and post-vaccination visits at Day 11, and Day 29 telephone contacts will be made on Day 91 and 181.
- Historical Control: Adults Aged 18-45: This arm consists of historical data from Vaxchora vaccine subjects from study PXVX-VC-200-004. The data was included in study PXVX-VC-200-005 as a comparator bridging population for the Day 11 seroconversion. NCT02094586, PubMed ID: 29317118
- Total: Total of all reporting groups
Arm/Group | PXVX0200 in Older Adults | Placebo in Older Adults | Historical Control: Adults Aged 18-45 | Total
Number analyzed (Participants) | 299 | 99 | 2688 | 3086
Age, Categorical [Count of Participants; unit: Participants]
  Between 46-64 years (inclusive): <=18 years | 0 | 0 | 0 | 0
  Between 46-64 years (inclusive): Between 18 and 65 years | 299 | 99 | 2688 | 3086
  Between 46-64 years (inclusive): >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (4.99) | 54.1 (5.20) | 30.0 (7.8) | 33.1 (NA) — Mean and standard deviation were not calculated for the total population as the historical control was not part of the original analysis of baseline characteristics. The historical control population is solely for comparison of immunogenicity variables in adults to older adults. Measures of dispersion of baseline characteristics across both populations is not applicable.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 52 | 1482 | 1698
  Male | 135 | 47 | 1206 | 1388
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 11 | 18
  Asian | 0 | 2 | 56 | 58
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 8 | 9
  Black or African American | 68 | 19 | 671 | 758
  White | 221 | 77 | 1855 | 2153
  More than one race | 2 | 0 | 50 | 52
  Unknown or Not Reported | 1 | 0 | 37 | 38
Region of Enrollment [Number; unit: participants]
  United States | 299 | 99 | 2341 | 2739
  Australia | 0 | 0 | 347 | 347

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate at Day 11
Description: The seroconversion rate is defined as the percentage of subjects with a 4-fold or greater rise over baseline Day 1 Serum Vibriocidal Antibody (SVA) titer against the classical Inaba biotype of V. cholerae at Day 11 following one dose of Vaxchora vaccine. The hypothesis was that the seroconversion rate would be non-inferior to the seroconversion rate at Day 11 in adults between the ages of 18 and 45 years.
Time Frame: Day 11
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | PXVX0200 in Older Adults | Historical Control: Adults Aged 18-45
Number analyzed (Participants) | 291 | 2687
% of participants | 90.4 [86.4 to 93.5] | 93.5 [92.5 to 94.4]
Statistical Analysis 1: Comparison: PXVX0200 in Older Adults vs Historical Control: Adults Aged 18-45; Test type: Non-Inferiority — The lower limit of the two sided 95% Wald CI on the difference in seroconversion rate was estimated by inverting a Z test with pooled variance. The lower limit of the CI had be greater than -10 percentage points to prove non-inferiority. The lower bound of the CI on the older adults serconversion rate was required to exceed 70%; Risk Difference (RD) = -3.1, 95% CI 2-sided [-6.7 to 0.4]

2. Secondary Outcome: Geometric Mean Titer (GMT)
Description: The Day 11 vibriocidal GMTs were compared between older and younger adults.
Time Frame: Day 11
Population: IEP
Measure: Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | PXVX0200 in Older Adults | Historical Control: Adults Aged 18-45 | Placebo in Older Adults
Number analyzed (Participants) | 291 | 2688 | 99
Geometric Mean Titer | 4282 [3344 to 5484] | 9688 [9067 to 10351] | 44 [36 to 56]
Statistical Analysis 1: Comparison: PXVX0200 in Older Adults vs Historical Control: Adults Aged 18-45; Test type: Other; Geometric Mean Ratio (GMR) = 0.44, 95% CI 2-sided [0.34 to 0.57]

3. Other Pre Specified Outcome: Cumulative Seroconversion Through Day 29 Compared to Day 11 for Younger Adults
Description: The cumulative seroconversion through Day 29 for older adults was compared to the Day 11 seroconversion for the younger adults aged 18 - 45 yrs. Seroconversion is defined as a 4-fold rise in antibody titer relative to baseline values.
Time Frame: Day 29
Population: IEP
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | PXVX0200 in Older Adults | Historical Control: Adults Aged 18-45 | Placebo in Older Adults
Number analyzed (Participants) | 291 | 2687 | 99
% of participants | 94.2 [90.8 to 96.6] | 93.5 [92.5 to 94.4] | 1.0 [0.0 to 5.5]
Statistical Analysis 1: Comparison: PXVX0200 in Older Adults vs Historical Control: Adults Aged 18-45; Test type: Non-Inferiority — Analysis for information only. No non-inferiority margin specified; Risk Difference (RD) = 0.6, 95% CI 2-sided [-2.2 to 3.5]

4. Other Pre Specified Outcome: Mean Fold Change in Vibriocidal Antibody Titer Between Day 1 and Day 11
Description: The mean log2 fold change between Day 1 and Day 11 in classical Inaba vibriocidal antibody titer attained by older adults was compared to the younger adults aged 18 - 45 yrs.
Time Frame: Day 11
Population: IEP. Placebo was not included in this additional bridging analysis as increase in SVA titer from Day 1 to 11 is not applicable for placebo subjects.
Measure: Mean (95% Confidence Interval); unit: Fold Change in Titer from Day 1
Arm/Group | PXVX0200 in Older Adults | Historical Control: Adults Aged 18-45
Number analyzed (Participants) | 291 | 2687
Fold Change in Titer from Day 1 | 6.6 [6.2 to 7.0] | 7.1 [7.0 to 7.3]
Statistical Analysis 1: Comparison: PXVX0200 in Older Adults vs Historical Control: Adults Aged 18-45; Test type: Non-Inferiority — Analysis for information only. No non-inferiority margin specified; p = 0.0062, t-test, 2 sided

5. Other Pre Specified Outcome: Seroconversion Against Other V. Cholerae Biotypes/Serotypes
Description: Seroconversion of the vibriocidal antibody response against 4 V. cholerae biotypes/serotypes - classical Inaba, El Tor Inaba, classical Ogawa and El Tor Ogawa was assessed.
Time Frame: Day 11
Population: IEP. The Historical Control population is not included as testing against these other biotypes/serotypes was not included in that study.
Measure: Mean (95% Confidence Interval); unit: % of participants
Arm/Group | PXVX0200 in Older Adults | Placebo in Older Adults
Number analyzed (Participants) | 291 | 99
% of participants
  Classical Inaba | 90.4 [86.4 to 93.5] | 0 [0.0 to 3.7]
  El Tor Inaba | 91.0 [87.1 to 94.1] | 5.1 [1.7 to 11.4]
  Classical Ogawa | 73.2 [67.7 to 78.2] | 2.0 [0.2 to 7.1]
  El Tor Ogawa | 71.4 [65.8 to 76.5] | 6.1 [2.3 to 12.7]

6. Other Pre Specified Outcome: Anti-CT Antibody Response in Older Adults
Description: The seroconversion of anti-Cholera Toxin (CT) antibody response in older adults was assessed.
  Seroconversion is defined as a 4-fold rise in anti-CT antibody titer relative to baseline values.
Time Frame: Day 11
Population: Immune Sub-Study Population. The Historical Control population is not included as anti-CT levels were not assessed in that study.
Measure: Mean (95% Confidence Interval); unit: % of participants
Arm/Group | PXVX0200 in Older Adults | Placebo in Older Adults
Number analyzed (Participants) | 36 | 9
% of participants | 55.6 [38.1 to 72.1] | 0 [0.0 to 33.6]

ADVERSE EVENTS:
Time Frame: Adverse event monitoring for this study will begin post-vaccination on Day 1 and will continue through Day 29 for all adverse events and the End-of-Study visit (Day 181) for serious adverse events. In order to fulfill safety reporting obligations, the Investigator should promptly report any SAEs resulting from study participation through the Day 181 visit.
Description: The Historical Control population is not included in this section as comparisons were not specified to be conducted in the protocol.
  Adverse events are reported for the safety population comprised of all randomized subjects who received either PXVX0200 or placebo.
Arm/Group | PXVX0200 in Older Adults | Placebo in Older Adults
All-Cause Mortality (participants affected / at risk) | 0/296 | 0/99
Serious Adverse Events (participants affected / at risk) | 3/296 | 0/99
Other Adverse Events (participants affected / at risk) | 37/296 | 11/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PXVX0200 in Older Adults (N=296) | Placebo in Older Adults (N=99)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PXVX0200 in Older Adults (N=296) | Placebo in Older Adults (N=99)
Fatigue (General disorders) | 11 | 3
Back Pain (Nervous system disorders) | 6 | 2
Decreased Appetite (Gastrointestinal disorders) | 5 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes